CLINICAL TRIAL: NCT01778907
Title: Effects and Cost-Effectiveness of Pharmacogenetic Screening Among Elderly Starters With Antidepressants: A Pragmatic Randomized Controlled Trial
Brief Title: Cytochrome P450-2D6 Screening Among Elderly Using Antidepressants (CYSCE)
Acronym: CYSCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Prof. Dr. Bob Wilffert, Prof. Dr. Bob Wilffert, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RUG11003
Record Dates: First submitted 2013-01-22; First posted 2013-01-29 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Depression; Depressive Disorder; Poor Metabolizer Due to Cytochrome P450 CYP2D6 Variant; Intermediate Metabolizer Due to Cytochrome P450 CYP2D6 Variant; Ultrarapid Metabolizer Due to Cytochrome P450 CYP2D6 Variant
Keywords: Pharmacogenetics; Depression; Depressive Disorder; Cytochrome P-450 CYP2D6; Antidepressive Agents, Tricyclic; Antidepressive Agents, Second-Generation; Poor Metabolizer Due to Cytochrome P450 CYP2D6 Variant; Intermediate Metabolizer Due to Cytochrome P450 CYP2D6 Variant; Ultrarapid Metabolizer Due to Cytochrome P450 CYP2D6 Variant; Multicenter studies
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal genotype- control (NG-C) (No Intervention): In the external control group, an advice for dose adaptation based on patients serum drug levels will be given to the physician according to current daily practice. Allocation to this arm is not based on randomization.
- Deviating genotype -control (DG-C) (No Intervention): In the internal control group, an advice for dose adaptation based on patients serum drug levels will be given to the physician according to current daily practice
- Deviating genotype (DG-I) (Experimental): In the intervention group, genotype information accompanied by a drug dosing advice will be given to the treating physician. Blood level of the drug will be communicated by a dedicated research team to the treating physician according to daily practice.
  Interventions: Other: Genotype information accompanied by a drug dosing advice

INTERVENTIONS:
Other: Genotype information accompanied by a drug dosing advice — Dosing advices for deviating genotypes (Poor Metabolizer, Intermediate Metabolizer, Ultrarapid Metabolizer)based on the guidelines of the Royal Dutch Pharmacists Association (KNMP).
  Arms: Deviating genotype (DG-I)

SUMMARY:
Depression is common among elderly with an estimated prevalence of 5%. Due to ageing the national burden will double in the coming decade. Antidepressants as TCAs and SSRIs are effective in reducing symptoms, especially in people with severe depression. To optimize treatment efficacy and reduce side effects, the Pharmacogenetics Working Group of the Royal Dutch Pharmacists Association developed guidelines for dose-adaptation, for instance for antidepressants such as nortriptyline and venlafaxine based on their main relevant genotype (CYP2D6) accompanied by Therapeutic Drug Monitoring. Such personalized drug dosing based on pharmacogenetic information at the start of therapy can speed up the titration phase of antidepressants to establish an adequate maintenance dose. However, pharmacogenetic screening programs are expensive and evidence on effects and costs of such a program among elderly antidepressant starters from randomized controlled studies is lacking. The investigators will conduct a pragmatic randomized controlled trial to determine the effects and costs of pharmacogenetic screening information to optimize drug dosing in depressed elderly patients who start with nortriptyline or venlafaxine.

Objective: The primary objective is to determine the effects of pharmacogenetic screening for CYP2D6 on the time to reach adequate blood levels as an accepted proxy for adequate treatment. Secondary objectives include adverse drug reactions and cost-effectiveness

Study design: pragmatic randomized controlled intervention study

DETAILED DESCRIPTION:
This study is a multicenter randomized controlled trial in which psychiatric elderly care centers participate in the Netherlands. Deviating genotypes are expected to be found in ~30% of the population, therefore the study consist out of two parts. First a basic study in which ~750 patients, starting with nortriptyline or venlafaxine will be genotyped to identify patients with deviating genotypes (Poor, Intermediate or Ultrarapid Metabolizers). Second in the main study 150 patients with a deviating genotype are randomly allocated to two study arms one with and one without information on the genotype. From the extensive metabolizers('normal'genotype) 75 patients are allocated to a third arm as an external control.

ELIGIBILITY:
Inclusion Criteria:

* Major depression according to DSM-IV (296.2x, 296.3x) criteria for which the treating psychiatrist decided to start drug treatment with either nortriptyline or venlafaxine.
* Competent to understand the informed consent procedure

Exclusion Criteria:

* Use of clinically relevant CYP2D6 inhibitors
* Use of clinically relevant CYP2D6 inducers
* Use of other drugs that affect plasma levels as co-medication
* Serious hepatic failure
* Patients for which drug treatment with venlafaxine is started and a GFR < 30 ml/min.
* Patients with the very rare genotype: Intermediate Metabolizer with duplications (IMDUP).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Serum drug levels of nortriptyline or venlafaxine | After 2, 4 and 6 weeks treatment started, after the 6th week sampling continues every 2 weeks untill adequate serum drug level is reached with an expected average of 8 weeks
  Serum drug levels will be assessed by 'dried blood spot' analysis, blood will be obtained by a fingerprick.
  Adequate serum drug levels is defined as: serum drug levels within the therapeutic window (for nortriptyline 50-150 µg/L, for venlafaxine 200-400 µg/L in combination with stable drug dosing for at least 3 weeks.

SECONDARY OUTCOMES:
Adverse drug events Questionnaire | At start of treatment and from that moment on, every 2 weeks untill adequate drug serum levels are reached with an expected average of 8 weeks
  Adverse drug events will be assessed by a self-reported questionnaire (ASEC). Two different questionnaires will be used, one for the side-effects of venlafaxine and another one for nortriptyline. Both are based one the ASEC questionnaire.
Quality of life questionnaire | After 2, 4 and 6 weeks treatment started and if adequate serum drug levels are not reached in 6 weeks, every 2 weeks, untill adequate serum drug levels are reached with an expected average of 8 weeks
  Quality of life will be assessed by the EQ5D questionnaire. This information will also be used for a cost-effectiveness analysis.
Productivity Questionnaire | After 2, 4 and 6 weeks treatment started and if adequate serum drug levels are not reached in 6 weeks, every 2 weeks, untill adequate serum drug levels are reached with an expected average of 8 weeks
  Effects on productivity by means of the Short Form-Health and Labour Questionnaire, part Labour. This information will also be used for a cost-effectiveness analysis.
Self reported Severity of depression Questionnaire | After 2, 4 and 6 weeks treatment started and if adequate serum drug levels are not reached in 6 weeks, every 2 weeks, untill adequate serum drug levels are reached with an expected average of 8 weeks
  Severity of depression by means of the QIDS-SR.
Drug use | At inclusion, after 2, 4 and 6 weeks after inclusion and if adequate serum drug levels are not reached in 6 weeks, every 2 weeks, untill adequate serum drug level is reached with an expected average of 8 weeks
  Drug use, including exact dosing and duration of prescription will be assessed by self reported drug use by the patient. This information will also be used for a cost-effectiveness analysis.
Data on health care associated resource use | After 2, 4 and 6 weeks treatment started and if adequate serum drug levels are not reached in 6 weeks, every 2 weeks, untill adequate serum drug levels are reached with an expected average of 8 weeks
  Data on health care associated resource use (e.g. visits to the specific specialists including diagnoses; drug use including exact dosing and durations of prescriptions; hospitalizations, inclusive exact intensities of care; and lab values if relevant). This information will also be used for a cost-effectiveness analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Bob Wilffert, Prof. Dr., Principal Investigator — University of Groningen; Eelko Hak, Prof. Dr., Principal Investigator — University of Groningen
Locations (11):
- Netherlands (11):
  - GGZ WNB, Halsteren, North Brabant
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Reinier van Arkel groep, 's-Hertogenbosch
  - GGz inGeest, Amsterdam
  - GGZ Centraal, Ermelo
  - Lentis, Groningen
  - University Medical Centre Groningen, Groningen
  - GGZ-NHN, Heiloo
  - GGZ Friesland, Leeuwarden
  - Parnassia, The Hague
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Berm EJ, Hak E, Postma M, Boshuisen M, Breuning L, Brouwers JR, Dhondt T, Jansen PA, Kok RM, Maring JG, van Marum R, Mulder H, Voshaar RC, Risselada AJ, Venema H, Vleugel L, Wilffert B. Effects and cost-effectiveness of pharmacogenetic screening for CYP2D6 among older adults starting therapy with nortriptyline or venlafaxine: study protocol for a pragmatic randomized controlled trial (CYSCEtrial). Trials. 2015 Jan 31;16:37. doi: 10.1186/s13063-015-0561-0. PMID 25636328
- [Derived] Berm EJ, Brummel-Mulder E, Paardekooper J, Hak E, Wilffert B, Maring JG. Determination of venlafaxine and O-desmethylvenlafaxine in dried blood spots for TDM purposes, using LC-MS/MS. Anal Bioanal Chem. 2014 Apr;406(9-10):2349-53. doi: 10.1007/s00216-014-7619-9. Epub 2014 Feb 4. PMID 24493333